CLINICAL TRIAL: NCT06245811
Title: Evaluation of the Relationship Between Hyperemesis Gravidarum (HEG) With Platelet Crit (PCT), Haemoglobin to Red Cell Distribution Width Ratio (HRR) and Neutrophil to Lymphocyte Ratio (NLR).
Brief Title: Inflammation Markers in Hyperemesis Gravidarum
Status: Completed | Type: Observational
Sponsor: Izzet Celegen (Other)
Responsible Party: Sponsor-Investigator, Izzet Celegen, Assistant professor, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Other Study IDs: UCKAN001
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Hyperemesis Gravidarum
Keywords: Hyperemesis gravidarum; Platelet criterion (PCT); Hemoglobin/red cell distribution width ratio (HRR); Neutrophil/lymphocyte ratio (NLR)
MeSH Terms: conditions — Hyperemesis Gravidarum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the relationship between the severity of hyperemesis gravidarum (HEG) disease and subclinical inflammatory factors such as Platelet Crit (PCT), Hemoglobin/red cell distribution width ratio (HRR), Neutrophil/lymphocyte ratio (NLR), was investigated.

DETAILED DESCRIPTION:
A total of 215 pregnant women, 102 with hyperemesis gravidarum and 113 healthy pregnant women, were included in the study. HEG patients were divided into three groups according to the modified PUQE classification: mild (n=38), moderate (n=32) and severe (n=32).

In our study, we proposed using a new prognostic marker for HEG patients. We think that our study will be a source for future studies on HEG.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women over 18 years of age
* 5-16 weeks of gestation.

Exclusion Criteria:

Smoking, urinary tract infections, previously diagnosed psychological disorders, gastrointestinal disorders, multiple pregnancies, eating disorders, thyroid disorders, inflammatory disease, pregnancy with assisted fertilization technique.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Healthy pregnant women over 18 years of age, 5-16 weeks of gestation.
Study Population: A total of 213 pregnant women, including 102 pregnant women with hyperemesis gravidarum and 113 healthy pregnant women between 5-16 weeks of age, were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
The Pregnancy Unique Quantification of Emesis/Stomach scoring system | 2 months
  1: Weight loss of 5% or more since the beginning of pregnancy 2: Vomiting at least three times a day 3: A ketonuria value of +1 or higher on a urinalysis test

SECONDARY OUTCOMES:
Body mass index | 2 months
  (BMI) (kg/m2) was obtained by dividing body weight (kg) by height (m2) squared

CONTACTS AND LOCATIONS:
Overall Officials: Kazım Uçkan, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Yuzuncu Yil University, Faculty of Medicine, Van, Turkey (Türkiye)